CLINICAL TRIAL: NCT04869397
Title: Treatment of Respiratory Complications Associated With COVID-19 Infection Using Wharton's Jelly (WJ)-Umbilical Cord (UC) Mesenchymal Stromal Cells (ProTrans®): a Randomized Phase II Controlled Clinical Trial
Brief Title: Treatment of Respiratory Complications Associated With COVID-19 Using Umbilical Cord Mesenchymal Stromal Cells
Acronym: ProTrans19+
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB advised discontinuing the study prematurely because recruitment goals were not achieved.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Ines Colmegna, Senior Researcher, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-6954
Record Dates: First submitted 2021-04-29; First posted 2021-05-03 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Covid19
Keywords: mesenchymal stromal cells; wharton's jelly; respiratory complication; biologics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic Wharton's jelly-MSCs (WJ-MSC) (Experimental): Intravenous administration, 1 dose, for 20 minutes
  Interventions: Biological: Allogeneic Wharton's jelly-MSCs (WJ-MSC)
- Placebo (Placebo Comparator): Intravenous administration, 1 dose, for 20 minutes
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Allogeneic Wharton's jelly-MSCs (WJ-MSC) — The product is provided cryopreserved by NextCell Pharma. The cells are frozen in cryobags at a concentration of 2 × 107 cells/ml in 5% Human Serum Albumin (HSA) and 10% dimethylsulfoxide (DMSO). One cryobag contains one dose. The bags are frozen in a controlled rate freezer and directly transferred to -190 ºC for storage until the time of infusion.
  Cryobags are thawed at bedside and diluted in 100 ml of saline prior to administration. Cells will be delivered at a rate of 5 million cells per minute over a total of 20 minutes.
  Other Names: Protrans
  Arms: Allogeneic Wharton's jelly-MSCs (WJ-MSC)
Other: Placebo — Sodium chloride buffer supplemented with 5% HSA and 10% DMSO same volume and mode of administration as treatment group
  Arms: Placebo

SUMMARY:
This is a randomized phase II placebo controlled clinical trial. Active arm: Allogeneic Wharton's jelly derived MSCs (WJ-MSCs). Both groups will receive standard of care treatment for COVID (e.g. dexamethasone)

DETAILED DESCRIPTION:
Allogeneic Wharton's jelly-MSCs (WJ-MSC) will be provided by NextCell Pharma under the commercial name of ProTrans®. ProTrans® will be administered at a fixed dose of 100 million cells per patient in a single infusion at bedside.

Placebo: Sodium chloride buffer supplemented with 5% HSA and 10% DMSO same volume and mode of administration as treatment group (NextCell Pharma).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years-old or older
* Laboratory-confirmed SARS-CoV-2 infection determined by reverse-transcription polymerase chain reaction (RT-PCR) prior to randomization
* Hospitalized patients
* Severe COVID-19 pneumonia defined as patients who cannot saturate > 96% on 4 L/min but are NOT on "non-invasive" ventilation nor invasive mechanical ventilation nor Extracorporeal membrane oxygenation (ECMO). Patients on high flow would be eligible if they receive treatment in a non-critical care unit only.
* Use of contraception or acceptable birth control for the duration of the study in women of childbearing potential
* Provision of written or verbal informed consent by the patient or designated substitute decision maker

Exclusion Criteria:

* Inability to provide informed consent
* Patients expected to survive less than 24 hours
* Advanced directives of patient's wishes to refuse intubation.
* Patients on mechanical ventilation
* Pregnant women [pregnancy defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotrophin (hCG) laboratory test]
* Breastfeeding
* Weight > 100 kg or < 50 kg
* Cancer not in remission or active serious illness unrelated to COVID-19.
* Any of the following laboratory results at screening: Absolute neutrophil count (ANC) ≤ 1.0 x 109/L, Platelets (PLT) < 50 G /L, Alanine transaminase (ALT) or Aspartate transaminase (AST) > 5N, eGFR < 30 mL/min
* Current documented bacterial infection
* Known infection with Human immunodeficiency virus, Treponema pallidum, Hepatitis B antigen (serology consistent with previous vaccination and a history of vaccination is acceptable) or Hepatitis C
* On-going therapy against tuberculosis, or exposed to tuberculosis or have travelled in areas with high risk of tuberculosis or mycosis within the last 3 months
* Known allergies to a component of the ProTrans® product
* Pre-existing chronic respiratory diseases requiring long-term oxygen therapy or severe pulmonary hypertension (PAPS >30 mm HG) or pulmonary fibrosis
* Pre-existing cirrhosis with basal Child and Pugh of C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Composite endpoint | at 15 days after intervention
  rate of use of mechanical ventilation (i.e. need for intubation) or death

SECONDARY OUTCOMES:
Clinical status evaluation assessed by the 9-point ordinal scale | day 7, 15 and 30
  Score 0. No clinical or virological evidence of infection. 1. No limitations of activities. 2. Ambulatory, limitation of activities. 3. Hospitalized, not requiring supplemental oxygen. 4. Hospitalized, requiring supplemental oxygen. 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices. 6. Hospitalized, intubated and on mechanical ventilation. 7. Hospitalized, ventilation + additional organ support - pressors, RRT, ECMO, 8. Death
Survival | day 7, 15 and 30
  Rate of patients alive at Day 7, Day 15 and Day 30
Time to clinical improvement assessed by the 9-point ordinal scale | time from randomization to either an improvement of 1 point on the 9-point ordinal scale or discharge from hospital
  Score 0. No clinical or virological evidence of infection. 1. No limitations of activities. 2. Ambulatory, limitation of activities. 3. Hospitalized, not requiring supplemental oxygen. 4. Hospitalized, requiring supplemental oxygen. 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices. 6. Hospitalized, intubated and on mechanical ventilation. 7. Hospitalized, ventilation + additional organ support - pressors, RRT (Renal Replacement Therapy), ECMO, 8. Death
Duration of hospitalization and ICU stay | From enrolment to discharge or ICU transfer or death
  Length of hospitalization and ICU stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Ines Colmegna, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada